CLINICAL TRIAL: NCT01807468
Title: Haploidentical Stem Cell Transplantation Followed by NK Cell Infusion in Patients With High-risk Solid Tumors Who Failed Autologous Stem Cell Transplantation
Brief Title: Haploidentical Stem Cell Transplantation and NK Cell Therapy in Patients With High-risk Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KiWoong Sung, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0113061
Record Dates: First submitted 2013-02-26; First posted 2013-03-08 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Neuroblastoma; Ewing Sarcoma; Rhabdomyosarcoma; Osteosarcoma; Soft Tissue Sarcoma
Keywords: haploidentical stem cell transplantation; natural killer cell therapy; pediatric solid tumor
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing; Rhabdomyosarcoma; Osteosarcoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HaploSC+NK (Experimental)
  Interventions: Procedure: haploidentical stem cell transplantation and NK cell therapy

INTERVENTIONS:
Procedure: haploidentical stem cell transplantation and NK cell therapy

SUMMARY:
To evaluate feasibility and efficacy of haploidentical stem cell transplantation in patients with high-risk solid tumors who failed after tandem high-dose chemotherapy and autologous stem cell transplantation.

To evaluate feasibility and efficacy of NK cell infusion after haploidentical stem cell transplantation in patients with high-risk solid tumors who failed after tandem high-dose chemotherapy and autologous stem cell transplantation.

DETAILED DESCRIPTION:
HaploSCT following reduced-intensity conditioning (RIC) regimen will be performed in patients with high-risk solid tumors. Both parents will be evaluated for their KIR genotype and phenotype and the one with the greatest degree of KIR-L mismatch with the patient will be selected as the donor. In addition, ex-vivo expanded NK cells derived from the donor will then be administered after haploSCT to increase the GVT effect. Low-dose IL-2 will be given after expanded NK cell infusion to enhance NK cell alloreactivity.

ELIGIBILITY:
Inclusion Criteria:

* age < 21 years old
* Patients with high-risk solid tumors who failed prior HDCT/autoSCT
* Patients with a suitable haploidentical donor
* High-risk solid tumors include high-risk neuroblastoma, metastatic or relapsed Ewing sarcoma, relapsed osteosarcoma, high-risk brain tumors, relapsed germ cell tumors, relapsed soft tissue sarcoma, relapsed rhabdomyosarcoma, and etc.
* stable disease with salvage chemotherapy after relapse

Exclusion Criteria:

* organ dysfunction(NCI common toxicity criteria grade > 2)
* progression of disease despite salvage chemotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of study patients with adverse events as a measure of safety of haploidentical stem cell transplantation and NK cell infusion | within 30 days after transplantation

SECONDARY OUTCOMES:
event-free survival and overall survival | 3 years after transplantation
  efficacy of haploidentical stem cell transplantation and NK cell infusion in patients with high-risk solid tumors

OTHER OUTCOMES:
number of patients developing GVHD | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, MD, PhD, Principal Investigator — Department of Pediatrics, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea